CLINICAL TRIAL: NCT03251781
Title: Determination of Minimal Important Difference for the Glittre-ADL Test and London Chest Activity of Daily Living Scale in Patients With COPD
Brief Title: Minimal Important Difference for the Glittre-ADL Test and London Chest Activity of Daily Living Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Prof. Dra. Anamaria Fleig Mayer, Principal Investigator, University of the State of Santa Catarina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 222/2011; 063053/2014 (Other: Universidade Federal de Ciências da Saúde de Porto Alegre)
Record Dates: First submitted 2017-07-28; First posted 2017-08-16 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Minimal Clinically Important Difference; Exercise Test; Rehabilitation; Disability Evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Pulmonary Rehabilitation
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Pulmonary rehabilitation program (PRP) was conducted according to the guidelines of the American Thoracic Society/European Respiratory Society (Nici et al., 2006; Spruit et al., 2013). Physical training was conducted over 24 sessions supervised, three times a week. The program included aerobic training in treadmill (with 30 min load determined by the dyspnea sensation - 4 to 6 on the modified Borg scale) and localized training for upper limbs with free weights or elastic bands (movements performed based on the proprioceptive neuromuscular facilitation diagonals, performed in two series, lasting two minutes each) and lower limbs (quadriceps and triceps sural) with free weights and/or in the bodybuilding station.

SUMMARY:
Background: The ability to perform activities of daily living (ADL) in patients with chronic obstructive pulmonary disease is often impaired. Glittre-ADL Test has been used to assess limitations in ADL, and it seems to be responsive to intervention. However, the minimal detectable change for Glittre-ADL Test remains unknown. Design: Non-controlled before and after study. Setting: The study will be conducted in an outpatient pulmonary rehabilitation program in Florianopolis, Brazil. Subjects: Patients with COPD (GOLD II-IV). Interventions: Pulmonary rehabilitation program based on physical training, conducted over 24 sessions supervised, three times a week, including aerobic training in treadmill and localized training for upper limbs and lower limbs. Main measures: Glittre ADL-Test performance, six-minute walk test performance, London Chest Activity of Daily Living score, Modified Medical Research Council score, COPD Assessment Test score, Saint George Respiratory Questionnaire score before and after the pulmonary rehabilitation program.

DETAILED DESCRIPTION:
Assigned Interventions: Pulmonary rehabilitation program (PRP) was conducted according to the guidelines of the American Thoracic Society/European Respiratory Society (ATS/ERS). Physical training was conducted over 24 sessions supervised, three times a week. The program included aerobic training in treadmill (with 30 min load determined by the dyspnea sensation - 4 to 6 on the modified Borg scale) and localized training for upper limbs with free weights or elastic bands (movements performed based on the proprioceptive neuromuscular facilitation diagonals, performed in two series, lasting two minutes each) and lower limbs (quadriceps and triceps sural) with free weights and/or in the bodybuilding station .

Pulmonary function test: Spirometry will be performed before the PRP, and it will be in accordance with ATS/ERS standards in order to provide the level of pulmonary obstruction and severity of disease. The predicted values will be calculated with the equations derived from Brazilian population.

Glittre-ADL Test: The patients will be instructed to complete five laps on the follow circuit as quickly as possible: from a sitting position, the subject stands up and walks along a flat 10-m long course, in the middle of which there is a two-step ladder (each step 17 cm high x 27 cm deep) to be climbed; after completing the 10 m, the subject faces a shelf containing three 1-kg objects positioned on the top shelf (shoulder height) and moves them one by one to the bottom shelf (waist height) and then to the floor; the objects are then returned to the bottom shelf and finally to the top shelf again; the subject walks back, climbing up and down the steps, until reaching the starting point (chair), sits down and immediately begins the next lap. The subjects carry a weighted backpack (2.5 kg for women, 5.0 kg for men). Two Glittre-ADL Tests will be conducted before and after the PRP.

Six minute walk test (6MWT): The patients will be instructed to walk in order to perform the largest distance during six minutes. The walking speed will be selected by the patient, according to the guidelines of the ATS. Two 6MWTs will be conducted before and after the PRP.

London Chest Activity of Daily Living scale: Patients will be asked about their perception of limitation in activities of daily living, using the London Chest Activity of Daily Living scale (LCADL) before and after the PRP.

Modified Medical Research Council scale: Patients will be asked about their perception of dyspnea, using the modified Medical Research Council scale before and after the PRP.

Saint George Respiratory Questionnaire: Patients will be asked about their perception of health-related quality of life, using the Saint George Respiratory Questionnaire before and after the PRP.

COPD Assessment Test (CAT): Patients will be asked about their perception of the impact of COPD (cough, sputum, dyspnea, and chest tightness) on health status, using CAT before and after the PRP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD confirmed by spirometry (COPD GOLD stages II, III and IV)
* Absence of change in respiratory symptoms in the past four weeks
* No hospital admission in the past 12 weeks
* Age between 40 and 80 years old

Exclusion Criteria:

* Any other disease or health condition that could compromise the test´s execution or physical training
* Participation in pulmonary rehabilitation program completed in the last six months
* Interruption of pulmonary rehabilitation program for any reason
* Current smoking or its cessation in less than six months
* Any change in symptoms during the study protocol assessments

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Glittre ADL-Test | The change in the Glittre ADL-test performance from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in Glittre ADL-Test performance
London Chest Activity of Daily Living | The change in the London Chest Activity of Daily Living score from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in London Chest Activity of Daily Living score

SECONDARY OUTCOMES:
Six-minute walking test | The change in the distance walked during the six-minute walking test from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in six-minute walking test performance
Modified Medical Research Council | The change in the Modified Medical Research Council score from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in Modified Medical Research Council score
COPD Assessment Test (CAT) | The change in the COPD Assessment Test (CAT) score from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in COPD Assessment Test (CAT) score
Saint George Respiratory Questionnaire (SGRQ) | The change in the Saint George Respiratory Questionnaire (SGRQ) score from baseline up to 24 pulmonary rehabilitation session (8 weeks of pulmonary rehabilitation).
  Change in Saint George Respiratory Questionnaire (SGRQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria F Mayer, PhD, Principal Investigator — University of the State of Santa Catarina
Locations (2):
- Brazil (2):
  - Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - University of the State of Santa Catarina, Florianópolis, Santa Catarina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Garrod R, Bestall JC, Paul EA, Wedzicha JA, Jones PW. Development and validation of a standardized measure of activity of daily living in patients with severe COPD: the London Chest Activity of Daily Living scale (LCADL). Respir Med. 2000 Jun;94(6):589-96. doi: 10.1053/rmed.2000.0786. PMID 10921765
- [Background] Carpes MF, Mayer AF, Simon KM, Jardim JR, Garrod R. The Brazilian Portuguese version of the London Chest Activity of Daily Living scale for use in patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Mar;34(3):143-51. doi: 10.1590/s1806-37132008000300004. English, Portuguese. PMID 18392462
- [Background] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Derived] Almeida Gulart A, de Araujo CLP, Bauer Munari A, Schneider BF, Dal Lago P, Mayer AF. Minimal important difference for London Chest Activity of Daily Living scale in patients with chronic obstructive pulmonary disease. Physiotherapy. 2020 Jun;107:28-35. doi: 10.1016/j.physio.2019.08.007. Epub 2019 Aug 9. PMID 32026830
- [Derived] Gulart AA, Araujo CLP, Munari AB, Santos KD, Karloh M, Foscarini BG, Dal Lago P, Mayer AF. The minimal important difference for Glittre-ADL test in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2020 Jan-Feb;24(1):54-60. doi: 10.1016/j.bjpt.2018.11.009. Epub 2018 Nov 20. PMID 30497829